CLINICAL TRIAL: NCT05010967
Title: Effect of High Intensity Interval Training Versus Yoga on Level of Pain, Catastrophizing and Quality of Life Among Females With Dysmenorrhea
Brief Title: Effect of HIIT VS Yoga on Level of Pain, Catastrophizing and QoL in Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01098 Areeba Aamir
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Primary Dysmenorrhea
Keywords: yoga; dysmenorrhea; Pain; catastrophizing; exercise
MeSH Terms: conditions — Dysmenorrhea; Pain; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental): High intensity interval training will be administered three days a week for 8 weeks. six series with 3 minutes rest period between series. For first 4 weeks the series would consist of 30 seconds of exercise and 30 seconds rest. exercises will consist of burpees, skipping, lunges, 1-legged squat, leg lever, push ups. for next four weeks the duration of exercise will be 45 seconds followed by 30 seconds recovery.
  Interventions: Other: High intensity interval training
- Yoga Training (Active Comparator): Yoga will be administered 3 days a week for 8 weeks. the session would be of 30-50 minutes with 5 minutes breathing followed by 15-35 minutes yoga and 10 minutes supine meditation. cat-cow stretch, child's pose, downward dog, plank, cobra pose will be used.
  Interventions: Other: Yoga Training

INTERVENTIONS:
Other: High intensity interval training — HIIT 3 times a week for 8 weeks. For week 1 to 4 , Warm up 5 minutes jogging in place, 6 series of 30 seconds Burpees, 30 seconds recovery, 30 seconds skipping, 30 seconds recovery, 30 seconds lunge, 30 seconds recovery, 30 seconds 1-legged squats, 30 seconds recovery, 30 second leg levers, 30 seconds recovery. the series will have 3 minutes rest in between. Cool down of 10 minutes with gentle stretches.
  For week 5 to 8 , Warm up 5 minutes jogging in place, 6 series of 45 seconds Burpees, 45 seconds recovery, 45 seconds skipping, 30 seconds recovery, 45 seconds lunge, 30 seconds recovery, 45 seconds 1-legged squats, 30 seconds recovery, 45 second leg levers, 30 seconds recovery. the series will have 3 minutes rest in between. Cool down of 10 minutes with gentle stretches.
  Arms: High intensity interval training
Other: Yoga Training — Yoga 3 times a week for 8 weeks. 30-50 minutes session, 5 minutes breathing, 15-35 minutes yoga poses (Cat-cow, child's pose, downward dog, plank, Cobra), followed by 10 minutes supine meditation.
  Arms: Yoga Training

SUMMARY:
This study is aimed at determining the effect of high intensity interval training VS yoga on pain, catastrophizing and quality of life among young females with dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea is defined as a pain experienced by females before or during menstruation and it is a common and important gynecological condition found in females of reproductive age that adversely affects their quality of life. The cause of PD is believed to be the excess release of prostaglandins during normal ovulation cycle.

The health care costs were altogether higher among females with dysmenorrhea compared with females who didn't experience the ill effects of this condition, and excess costs were essentially determined by outpatient care, so poses greater burden of disease than any other gynecological complaint. Females having more pain catastrophizing scores leads to increases chances of disability. Proper evidence behind HIIT training among females with primary dysmenorrhea is sparse and is based on different clinical experiences and a less number of studies with limited methodological design.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried Females with age 18-25 years
* Normal Menstrual cycles 21-35 days
* Primary Dysmenorrhea diagnosis made on the WaLIDD score
* WaLIDD score of 1- 7 (Mild to moderate dysmenorrhea)

Exclusion Criteria:

* History of regular exercise (3 times weekly for 30-45 min)
* Motor Disabilities ( ALS, Multiple sclerosis, Muscular dystrophy )
* Autoimmune conditions (RA, Hashimotos Thyroiditis)
* Chronic illnesses that might contraindicate physical exercise (asthma, epilepsy, migraine, anemia, complete heart block, acute congestive heart failure, unstable angina, and uncontrolled severe hypertension)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study is focused on females with dysmenorrhea.
Enrollment: 34 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 8th week
  changes from baseline The numeric pain rating scale (NPRS) is a 10 points scale on which, zero represent no pain, 1 to 3 represent mild pain, 4 to 7 represent moderate and pain score between 7 and 10 were considered to be a severe form of pain.[

SECONDARY OUTCOMES:
Pain catastrophizing | 8th week
  The 13-item scale measures the extent to which participants worry, amplify, and feel helpless about the experience of pain on a five-point (0-4) scale. Total scores range from 0 to 52, with higher scores indicating greater pain catastrophizing.
EQ-5D for quality of life | 8th week
  The EQ-5D is an acceptable, reliable and valid measure of quality of life. The EQ-5D, a standardized questionnaire consists of two parts: the first is the 'EQ-5D descriptive system' with five questions about several dimensions of HrQoL (mobility, self-care, daily activities, pain/discomfort and anxiety/depression). Each dimension can be rated at three levels: 'no problems', 'some problems' and 'major problems'. The responses to the five dimensions together lead to an aggregated index, the 'EQ-5D index', which corresponds to a health state. The second part of the scale is the 'EQ Visual Analogic Scale' (EQVAS) which is the respondent's own assessment of her overall health status on a thermometer-like visual scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Martinez E, Onieva-Zafra MD, Parra-Fernandez ML. Lifestyle and prevalence of dysmenorrhea among Spanish female university students. PLoS One. 2018 Aug 10;13(8):e0201894. doi: 10.1371/journal.pone.0201894. eCollection 2018. PMID 30096156
- [Background] Akiyama S, Tanaka E, Cristeau O, Onishi Y, Osuga Y. Evaluation of the treatment patterns and economic burden of dysmenorrhea in Japanese women, using a claims database. Clinicoecon Outcomes Res. 2017 May 22;9:295-306. doi: 10.2147/CEOR.S127760. eCollection 2017. PMID 28579813
- [Background] Hu Z, Tang L, Chen L, Kaminga AC, Xu H. Prevalence and Risk Factors Associated with Primary Dysmenorrhea among Chinese Female University Students: A Cross-sectional Study. J Pediatr Adolesc Gynecol. 2020 Feb;33(1):15-22. doi: 10.1016/j.jpag.2019.09.004. Epub 2019 Sep 17. PMID 31539615
- [Background] Aubry G, Panel P, Thiollier G, Huchon C, Fauconnier A. Measuring health-related quality of life in women with endometriosis: comparing the clinimetric properties of the Endometriosis Health Profile-5 (EHP-5) and the EuroQol-5D (EQ-5D). Hum Reprod. 2017 Jun 1;32(6):1258-1269. doi: 10.1093/humrep/dex057. PMID 28383700
- [Background] Durand H, Monahan K, McGuire BE. Prevalence and Impact of Dysmenorrhea Among University Students in Ireland. Pain Med. 2021 Dec 11;22(12):2835-2845. doi: 10.1093/pm/pnab122. PMID 33822197
- [Background] Yang NY, Kim SD. Effects of a Yoga Program on Menstrual Cramps and Menstrual Distress in Undergraduate Students with Primary Dysmenorrhea: A Single-Blind, Randomized Controlled Trial. J Altern Complement Med. 2016 Sep;22(9):732-8. doi: 10.1089/acm.2016.0058. Epub 2016 Jun 17. PMID 27315239
- [Background] Yonglitthipagon P, Muansiangsai S, Wongkhumngern W, Donpunha W, Chanavirut R, Siritaratiwat W, Mato L, Eungpinichpong W, Janyacharoen T. Effect of yoga on the menstrual pain, physical fitness, and quality of life of young women with primary dysmenorrhea. J Bodyw Mov Ther. 2017 Oct;21(4):840-846. doi: 10.1016/j.jbmt.2017.01.014. Epub 2017 Feb 7. PMID 29037637
- [Background] McGovern CE, Cheung C. Yoga and Quality of Life in Women with Primary Dysmenorrhea: A Systematic Review. J Midwifery Womens Health. 2018 Jul;63(4):470-482. doi: 10.1111/jmwh.12729. Epub 2018 Jun 14. PMID 29902363
- [Background] P. Guruprasad, Padmaja and Sharma, Urvashi and Palekar, Tushar and Pimpri, "Immediate Effect of Yoga Postures v/s Physiotherapy Exercises Along With KTaping on Pain in Dysmenorrhea," 2019.
- [Background] P. Prabhu, Shraddha and Nagrale, Sanket and Shyam, Ashok and Sancheti, "Effect of yogasanas on menstrual cramps in young adult females with primary dysmenorrhea," Int J Physiother Res, vol. 7, no. 4, pp. 3109--3112, 2019.
- [Background] Sperlich B, Wallmann-Sperlich B, Zinner C, Von Stauffenberg V, Losert H, Holmberg HC. Functional High-Intensity Circuit Training Improves Body Composition, Peak Oxygen Uptake, Strength, and Alters Certain Dimensions of Quality of Life in Overweight Women. Front Physiol. 2017 Apr 3;8:172. doi: 10.3389/fphys.2017.00172. eCollection 2017. PMID 28420999
- [Background] J. R. Rahimi, Niloofar, Effat Bambaiechi, "Comparison the effect of eight weeks high intensity interval and moderate continuous trainings on pain reductionand and blood levels of IL6 and TNF-α in woman with primary dysmenorrhea," Res. Med., vol. 41, no. 4, pp. 258--268, 2017
- [Background] Sperlich B, Hahn LS, Edel A, Behr T, Helmprobst J, Leppich R, Wallmann-Sperlich B, Holmberg HC. A 4-Week Intervention Involving Mobile-Based Daily 6-Minute Micro-Sessions of Functional High-Intensity Circuit Training Improves Strength and Quality of Life, but Not Cardio-Respiratory Fitness of Young Untrained Adults. Front Physiol. 2018 May 9;9:423. doi: 10.3389/fphys.2018.00423. eCollection 2018. PMID 29867519
- [Background] Kirmizigil B, Demiralp C. Effectiveness of functional exercises on pain and sleep quality in patients with primary dysmenorrhea: a randomized clinical trial. Arch Gynecol Obstet. 2020 Jul;302(1):153-163. doi: 10.1007/s00404-020-05579-2. Epub 2020 May 15. PMID 32415471
- [Background] Kannan P, Chapple CM, Miller D, Claydon-Mueller L, Baxter GD. Effectiveness of a treadmill-based aerobic exercise intervention on pain, daily functioning, and quality of life in women with primary dysmenorrhea: A randomized controlled trial. Contemp Clin Trials. 2019 Jun;81:80-86. doi: 10.1016/j.cct.2019.05.004. Epub 2019 May 7. PMID 31071464
- [Background] S. I. and others Aiyegbusi, Ayoola Ibifubara and Adeagbo, Caleb Adewunmi and Uwem-Umoh, "Comparative efficacy of core strengthening and stretching exercises on systemic and quality-of-life symptoms in adolescent college students with primary dysmenorrhea," New Niger. J. Clin. Res., vol. 9, no. 16, p. 59, 2020.
- [Background] Heidarimoghadam R, Abdolmaleki E, Kazemi F, Masoumi SZ, Khodakarami B, Mohammadi Y. The Effect of Exercise Plan Based on FITT Protocol on Primary Dysmenorrhea in Medical Students: A Clinical Trial Study. J Res Health Sci. 2019 Aug 24;19(3):e00456. PMID 31586377
- [Background] S. Atashak, Sirvan and Rashidi, "Effect of eight-week high-intensity interval training and ginger supplementation on primary dysmenorrhea in nonathletic female students," Iran. J. Obstet. Gynecol. Infertil., vol. 20, no. 12, pp. 23--31, 2018.
- [Background] T. N. Ouda, Khalil, Sameh Latif, "A study of the effect of heat application on relieving dysmenorrheal pain among young females," African J. Nurs. Midwifery, vol. 5, no. 6, pp. 727-735, 2017.
- [Background] B. S. M. Ameade, EP Kwuame, "Menstrual pain assessment: comparing verbal rating scale (VRS) with numerical rating scales (NRS) as pain measurement tools," 2016
- [Background] Chen CX, Carpenter JS, LaPradd M, Ofner S, Fortenberry JD. Perceived Ineffectiveness of Pharmacological Treatments for Dysmenorrhea. J Womens Health (Larchmt). 2021 Sep;30(9):1334-1343. doi: 10.1089/jwh.2020.8581. Epub 2020 Oct 7. PMID 33026968
- [Background] Rakhshaee Z. Effect of three yoga poses (cobra, cat and fish poses) in women with primary dysmenorrhea: a randomized clinical trial. J Pediatr Adolesc Gynecol. 2011 Aug;24(4):192-6. doi: 10.1016/j.jpag.2011.01.059. Epub 2011 Apr 21. PMID 21514190
- [Background] Tsai SY. Effect of Yoga Exercise on Premenstrual Symptoms among Female Employees in Taiwan. Int J Environ Res Public Health. 2016 Jul 16;13(7):721. doi: 10.3390/ijerph13070721. PMID 27438845